CLINICAL TRIAL: NCT03730779
Title: Normobaric Nocturnal Hyperoxia Therapy for Treating Ischemic-Related Retinal Conditions
Brief Title: Oxygen Therapy for Retinal Ischemia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Jorge Arroyo, Associate Professor of Ophthalmology, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Trials2018
Record Dates: First submitted 2018-11-02; First posted 2018-11-05 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Retinal Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- O2 recieving (Experimental): Patients who receive hyperoxia
  Interventions: Drug: Hyperoxia

INTERVENTIONS:
Drug: Hyperoxia — Patients will receive nocturnal normobaric hyperoxia therapy
  Other Names: Nocturnal normobaric hyperoxia

SUMMARY:
The investigators will be using nocturnal normobaric hyperoxia therapy in patients with diagnoses of conditions related to retinal ischemia.

DETAILED DESCRIPTION:
Patients who receive a diagnosis of a condition relate to retinal ischemia and who pass the eligibility criteria will receive an oxygen concentrator to use at home. They will report back in follow up monthly for three to six months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of retinal-ischemia related condition

Exclusion Criteria:

* Complicating other ocular condition
* History of smoking or lung conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | 6 months
  Best Corrected Visual Acuity as measured by ETDRS chart
Macula Edema | 6 months
  Amount of ME present, as measured by OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
If researchers wish to access IPD they may contact us with their request